CLINICAL TRIAL: NCT01628731
Title: Phase III Study of Furosemide Continuous Infusion Versus Ethacrynic Acid Continuous Infusion in Children Undergoing Cardiac Surgery: Randomized Double Blind Controlled Clinical Trial
Brief Title: Furosemide Versus Ethacrynic Acid in Children With Congenital Heart Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bambino Gesù Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Zaccaria Ricci, Medical Doctor, Research Fellow, Bambino Gesù Hospital and Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FUROCRYNIC trial-1; OBG DIURETICS (Other: Bambino Gesù Hospital RI)
Record Dates: First submitted 2012-06-24; First posted 2012-06-27 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Fluid Overload
Keywords: loop diuretics; fluid balance; urine output; acute renal dysfunction
MeSH Terms: conditions — Edema | interventions — Furosemide; Ethacrynic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- furosemide (Active Comparator): furosemide, 0.2 mg/kg/h up to 0.8 mg/kg/h for 72 hours
  Interventions: Drug: furosemide
- ethacryinic acid (Active Comparator): ethacrynic acid, 0.2 mg/kg/h up to 0.8 mg/kg/h for 72 hours
  Interventions: Drug: ethacrynic acid

INTERVENTIONS:
Drug: furosemide — furosemide, intravenous, continuous infusion, 0.2 mg/kg/h for 24 hours
  Other Names: lasix
  Arms: furosemide
Drug: ethacrynic acid — ethacrynic acid, intravenous, continuous infusion, 0.2 mg/kg/h for 24 hours
  Other Names: reomax
  Arms: ethacryinic acid

SUMMARY:
This study aims to verify if ethacrynic acid continuous infusion is superior to furosemide continuous infusion in total urine output production during the first 24 post operative hours.

DETAILED DESCRIPTION:
Diuretic therapy in children after open heart surgery is widely administered, though no evidence currently supports if an ideal drug or an ideal dosage can be recommended. Loop diuretics are the most effective drugs in terms of urine output production but may cause some collateral effects such as metabolic alkalosis, hypovolemia, hypokalemia, ototoxicity. Furthermore, some reports showed that loop diuretics usage can be associated with an increased risk of renal dysfunction and mortality. However, their use in children with signs of fluid overload, pulmonary edema or oliguria is mandatory and widely practiced.

Furosemide and ethacrynic acid are often prescribed and administered without any specific indication, basing on clinicians preferences.

No study so far, explored the hypothesis of which of these drugs is the most effective in terms of urine output production and safe in terms of renal function.

This study aims to verify if ethacrynic acid continuous infusion is superior to furosemide continuous infusion in total urine output production during the first 24 post operative hours.

ELIGIBILITY:
Inclusion Criteria:

* Children with congenital heart disease undergoing cardiac surgery
* intraoperative aortic cross clamp over 90 minutes or interventional catheterization procedures with post-operative inotrope score over 20
* sign of fluid retention after surgical procedures

Exclusion Criteria:

* Preoperative renal dysfunction
* Preoperative administration of more than 4mg/kg/die loop diuretics
* Need for renal replacement therapy at ICU admission
* Need for ECMO at ICU admission

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 2012-10; Primary Completion 2013-07 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Mean total urine output production in the first post-operative day | first 24 hours after Intensive Care Unit admission
  Verification of the superiority of ethacrynic acid compared with furosemide in improving patients' total urine output by at least 1 ml/kg/h in the first 24 post-operative hours

SECONDARY OUTCOMES:
Mean creatinine and NGAL values | first 72 hours after Intensive Care Unit admission
  Verification of the superiority of ethacrynic acid compared with furosemide in improving patients' renal function (asessed as creatinine, NGAL and pRIFLE score) in the first 72 post-operative hours

CONTACTS AND LOCATIONS:
Overall Officials: Zaccaria Ricci, MD, Principal Investigator — Bambino Gesù Hospital RI
Locations (1):
- Bambino Gesù Hospital, Rome, Italy

REFERENCES:
- [Background] Klinge JM, Scharf J, Hofbeck M, Gerling S, Bonakdar S, Singer H. Intermittent administration of furosemide versus continuous infusion in the postoperative management of children following open heart surgery. Intensive Care Med. 1997 Jun;23(6):693-7. doi: 10.1007/s001340050395. PMID 9255651
- [Background] van der Vorst MM, Ruys-Dudok van Heel I, Kist-van Holthe JE, den Hartigh J, Schoemaker RC, Cohen AF, Burggraaf J. Continuous intravenous furosemide in haemodynamically unstable children after cardiac surgery. Intensive Care Med. 2001 Apr;27(4):711-5. doi: 10.1007/s001340000819. PMID 11398698
- [Background] Bagshaw SM, Gibney RT, McAlister FA, Bellomo R. The SPARK Study: a phase II randomized blinded controlled trial of the effect of furosemide in critically ill patients with early acute kidney injury. Trials. 2010 May 11;11:50. doi: 10.1186/1745-6215-11-50. PMID 20459801
- [Derived] Ricci Z, Haiberger R, Pezzella C, Garisto C, Favia I, Cogo P. Furosemide versus ethacrynic acid in pediatric patients undergoing cardiac surgery: a randomized controlled trial. Crit Care. 2015 Jan 7;19(1):2. doi: 10.1186/s13054-014-0724-5. PMID 25563826